CLINICAL TRIAL: NCT05467241
Title: A Pilot Study to Assess the Feasibility of a Randomized Control Trial Employing a Single-arm Intervention, at a Single Institution, to Study the Effects of Combined Self-induced Therapeutic Tremors Plus Mindfulness on Symptoms of Chronic Pelvic Pain.
Brief Title: A Novel Therapeutic Approach to Treat Chronic Pelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee Graduate School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4818
Record Dates: First submitted 2021-09-07; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pelvic Pain
MeSH Terms: interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Combined Alternative Therapy: The novel combined alternative therapy that will be studied consists of self-induced therapeutic tremors (SITT) plus mindfulness. SITT is the intentional induction of the body's innate tremor mechanism to treat hyperarousal and muscle tension, which is characteristic of CPP. SITTs are thought to restore somatic and autonomic nervous system homeostasis, by discharging sympathetic arousal and down-regulating the autonomic nervous system. Previous work has shown that mindfulness training may improve symptoms of CPP, however there are no studies investigating the impact that the combination of mindfulness coupled with SITTs may have on the symptoms of CPP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self-induced therapeutic tremor (SITT) combined with mindfulness (Experimental): This arm will consist of self-induced therapeutic tremor (SITT) training combined with mindfulness training that is performed during a 60 minute session, 2 times per week, for 4 weeks.
  Self-induced therapeutic tremor (SITT) combined with mindfulness: SITT is a way to reduce stress by turning on a natural shaking response. This can calm the participant's body. It involves doing simple exercises. During SITT muscles will gently shake, and release built up stress. This shaking of muscles lets the participant's body physically let go of tension and stress. Mindfulness is the ability to be fully present in a moment so that the participant can focus on what the participant is sensing and feeling in the moment. It involves the acceptance of thoughts and feelings without judging them. Practicing mindfulness involves breathing methods, guided imagery, and other practices to relax the body and mind, help reduce stress, and not be overwhelmed.
  Interventions: Behavioral: Self-induced therapeutic tremor (SITT) combined with mindfulness

INTERVENTIONS:
Behavioral: Self-induced therapeutic tremor (SITT) combined with mindfulness — SITT is a way to reduce stress by turning on a natural shaking response. This can calm the participant's body. It involves doing simple exercises. The muscles will gently shake, and release built up stress. This shaking of the muscles lets the participant's body physically let go of tension and stress.
  Mindfulness is the ability to be fully present in a moment. This allows focus on what the participant is sensing and feeling in the moment. It involves the acceptance of thoughts and feelings without judging them.
  Practicing mindfulness involves breathing methods, guided imagery, and other practices to relax the body and mind, help reduce stress, and not be overwhelmed by what's going on around the participant.

SUMMARY:
To collect pilot data and assess the feasibility of a trial employing a single-arm intervention to study the effects of combined self-induced therapeutic tremors plus mindfulness on symptoms of chronic pelvic pain among women diagnosed with chronic pelvic pain.

DETAILED DESCRIPTION:
The estimated prevalence of chronic pelvic pain among women is 2-24%. The etiology of chronic pelvic pain is multifactorial making it very difficult to manage clinically. Evidenced-based therapies are limited and a multidisciplinary approach, including complementary and alternative medicine, to treat women with chronic pelvic pain may be the best approach. This study assess the feasibility of conducting randomized controlled trial with a single arm intervention to treat symptoms of chronic pelvis pain among women diagnosed with chronic pelvic pain. The intervention will consist of a novel combined alternative therapy intervention among women with chronic pelvic pain (self-induced therapeutic tremor plus mindfulness). This is a clinically significant project as lifestyle interventions to treat chronic pelvic pain are urgently needed, given the prevalence and the healthcare costs associated with chronic pelvic pain.

Study Objective: The primary purpose of this project is to collect pilot data and assess the feasibility of a single arm intervention trial to improve symptoms of CPP among women diagnosed with CPP.

Intervention Arm - Combined Alternative Therapy: The novel combined alternative therapy that will be studied consists of self-induced therapeutic tremors (SITT) plus mindfulness. SITT is the intentional induction of the body's innate tremor mechanism to treat hyperarousal and muscle tension, which is characteristic of CPP. SITTs are thought to restore somatic and autonomic nervous system homeostasis, by discharging sympathetic arousal and down-regulating the autonomic nervous system. Previous work has shown that mindfulness training may improve symptoms of CPP, however there are no studies investigating the impact that the combination of mindfulness coupled with SITTs may have on the symptoms of CPP.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age >18
* Physical requirements: be able to complete the intervention sessions
* Not seeking other therapeutic modalities, such as acupuncture, PT, during study duration
* Free from surgery for >3 months
* being treated clinically for chronic pelvic pain and related conditions
* CPP of 6 months or more (to be considered chronic)
* Availability to commit to the 4-week intervention (two 60-minute sessions per week at a specified time, for 4 weeks)
* Internet access and consistent access to phone/email/text communication

Exclusion Criteria:

* Pregnancy
* Illicit substance use (e.g. cocaine, methamphetamines, heroin, street drugs) - marijuana and CBD oil and related supplements will be considered on a case-by-case basis by the principal investigators
* Current psychiatric illness/social situation that would limit compliance with study requirements, as determined by the principal investigators

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the pilot trial | This will be assessed at the completion of the study, approximately 1-1.5 years after the study start.
  To determine feasibility, the investigators will assess if it is possible to recruit, enroll, and have complete follow-up with participants. If the recruitment goal is met and 80% compliance with study visit attendance is achieved, the trial will be classified as feasible (yes/no classification).

SECONDARY OUTCOMES:
Change in Physical Function | Pre- Program, Immediately Post-Program, and 1 Month Follow Up
  PROMIS-29 Profile v2.0 Questionnaire will be used to assess the domain of Physical Function. This domain is assessed with 4 questions. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, the values of all 4 questions are summed. The lowest value is 4 and the highest value is 20. These total raw scores are converted into T-scores using the appropriate tables in the appropriate appendix in the "PROMIS ADULT PROFILE INSTRUMENTS SCORING MANUAL." The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more of this concept being measured. For this domain specifically, a higher score is a better outcome.
  The change in T-score for this domain, across time, is assessed using repeated measures ANOVA.
Change in Anxiety | Pre- Program, Immediately Post-Program, and 1 Month Follow Up
  PROMIS-29 Profile v2.0 Questionnaire will be used to assess the domain of Anxiety. This domain is assessed with 4 questions. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, the values of all 4 questions are summed. The lowest value is 4 and the highest value is 20. These total raw scores are converted into T-scores using the appropriate tables in the appropriate appendix in the "PROMIS ADULT PROFILE INSTRUMENTS SCORING MANUAL." The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more of this concept being measured. For this domain specifically, a higher score is a worse outcome.
  The change in T-score for this domain, across time, is assessed using repeated measures ANOVA.
Change in Depression | Pre- Program, Immediately Post-Program, and 1 Month Follow Up
  PROMIS-29 Profile v2.0 Questionnaire will be used to assess the domain of Depression. This domain is assessed with 4 questions. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, the values of all 4 questions are summed. The lowest value is 4 and the highest value is 20. These total raw scores are converted into T-scores using the appropriate tables in the appropriate appendix in the "PROMIS ADULT PROFILE INSTRUMENTS SCORING MANUAL." The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more of this concept being measured. For this domain specifically, a higher score is a worse outcome.
  The change in T-score for this domain, across time, is assessed using repeated measures ANOVA.
Change in Fatigue | Pre- Program, Immediately Post-Program, and 1 Month Follow Up
  PROMIS-29 Profile v2.0 Questionnaire will be used to assess the domain of Fatigue. This domain is assessed with 4 questions. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, the values of all 4 questions are summed. The lowest value is 4 and the highest value is 20. These total raw scores are converted into T-scores using the appropriate tables in the appropriate appendix in the "PROMIS ADULT PROFILE INSTRUMENTS SCORING MANUAL." The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more of this concept being measured. For this domain specifically, a higher score is a worse outcome.
  The change in T-score for this domain, across time, is assessed using repeated measures ANOVA.
Change in Sleep Disturbance | Pre- Program, Immediately Post-Program, and 1 Month Follow Up
  PROMIS-29 Profile v2.0 Questionnaire will be used to assess the domain of Sleep Disturbance. This domain is assessed with 4 questions. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, the values of all 4 questions are summed. The lowest value is 4 and the highest value is 20. These total raw scores are converted into T-scores using the appropriate tables in the appropriate appendix in the "PROMIS ADULT PROFILE INSTRUMENTS SCORING MANUAL." The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more of this concept being measured. For this domain specifically, a higher score is a worse outcome.
  The change in T-score for this domain, across time, is assessed using repeated measures ANOVA.
Change in Ability to Participant in Social Roles and Activities | Pre- Program, Immediately Post-Program, and 1 Month Follow Up
  PROMIS-29 Profile v2.0 Questionnaire will be used to assess the domain of Ability to Participate in Social Roles and Activities. This domain is assessed with 4 questions. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, the values of all 4 questions are summed. The lowest value is 4 and the highest value is 20. These total raw scores are converted into T-scores using the appropriate tables in the appropriate appendix in the "PROMIS ADULT PROFILE INSTRUMENTS SCORING MANUAL." The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more of this concept being measured. For this domain specifically, a higher score is a better outcome.
  The change in T-score for this domain, across time, is assessed using repeated measures ANOVA.
Change in Pain Intensity | Pre- Program, Immediately Post-Program, and 1 Month Follow Up
  PROMIS-29 Profile v2.0 Questionnaire will be used to assess the domain of Pain Intensity. This domain is assessed with 4 questions. Each question has 5 response options ranging in value from 1 to 5. To find the total raw score, the values of all 4 questions are summed. The lowest value is 4 and the highest value is 20. These total raw scores are converted into T-scores using the appropriate tables in the appropriate appendix in the "PROMIS ADULT PROFILE INSTRUMENTS SCORING MANUAL." The T-score rescales the raw score into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. A higher score represents more of this concept being measured. For this domain specifically, a higher score is a worse outcome.
  The change in T-score for this domain, across time, is assessed using repeated measures ANOVA.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Tennessee Graduate School of Medicine, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No